CLINICAL TRIAL: NCT07120503
Title: A Phase 2 Randomized, Double-blind Placebo-Controlled Study to Evaluate the Pharmacokinetics, Immunogenicity, Safety and Efficacy of WIN378 in Adult Participants With Moderate or Severe Asthma
Brief Title: Study to Evaluate the Safety, Pharmacology and Efficacy of WIN378 in Adults With Moderate or Severe Asthma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Windward Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WB-2101; 2025-521391-58-00 (EU CTIS Number); U1111-1319-6369 (Other: UTN, World Health Organization (WHO))
Record Dates: First submitted 2025-07-25; First posted 2025-08-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Asthma (Diagnosis)
Keywords: Asthma; Moderate Asthma; Severe Asthma; Uncontrolled Asthma; Respiratory Diseases; Lung Diseases; Bronchial Diseases; Allergic Diseases
MeSH Terms: conditions — Asthma; Disease; Respiratory Tract Diseases; Lung Diseases; Bronchial Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- WIN378 (Experimental): WIN378 SC injections
  Interventions: Drug: WIN378
- Placebo (Experimental): Placebo SC Injections
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: WIN378 — WIN378 is a fully human, long-acting monoclonal antibody that binds to thymic stromal lymphopoietin (TSLP), blocking its activity and thereby reducing airway inflammation and improving asthma control over an extended dosing interval.
  Arms: WIN378
Drug: Placebo — A sham injection consisting of placebo to mask WIN378.
  Arms: Placebo

SUMMARY:
This study is trying to identify the right dose of a long-acting medicine called WIN378 for people with moderate or severe asthma. WIN378 blocks the action of a protein called TSLP which causes inflammation in the lung and may contribute to your asthma control and symptoms. The study will test how doses of WIN378 are handled by your body (pharmacokinetics) and assess the safety of the medicine and will assess markers of asthma inflammation in your breath and in your blood, lung function and asthma control (pharmacodynamics).

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled, dose-ranging study to evaluate the safety, tolerability, efficacy and pharmacokinetics of WIN378 in adult participants with moderate to severe asthma. Participants will continue their standard background asthma therapy according to GINA Steps 3-5. Eligible participants will be randomized to receive WIN378 or placebo administered subcutaneously over a 48-week treatment period, followed by a 12-week safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent Form
* Females that are not pregnant or breastfeeding with following condition: not a woman of childbearing potential or woman of childbearing potential using a highly effective contraception method
* Physician-diagnosis of asthma and documented evidence of airway reversibility during prior 24 months or during screening
* Airflow limitation as indicated by pre-BD FEV1 value of ≥ 30% and ≤ 90%, predicted at two visits at Screening
* Low, medium-, or high-dose ICS and ≥1 maintenance asthma controller medication (LABA/LTRA/LAMA/chromones/theophylline)

Exclusion Criteria:

* Participants with a known, pre-existing, clinically important lung condition other than asthma
* Active tuberculosis or treatment required for tuberculosis within 12 months
* Current or former smokers ≥10 pack years
* History of cancer
* Receipt of any marketed biologic agent within 4 months or 5 half-lives prior to screening; receipt of immunoglobulin or blood products within 30 days prior to screening or during the Screening Run-in period; receipt of any live or attenuated vaccines within 15 days prior to screening
* Helminth infection within 24 weeks prior to screening
* Use of immunosuppressive medication within 3 months prior to Screening Visit or during the Screening Run-in period
* Participants who are pregnant, lactating or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) during the study | Week 0 - Week 60
Number of participants with treatment-emergent serious adverse events (TESAEs) during the study | Week 0 - Week 60
Number of participants with abnormal vital signs during the study | Week 0 - Week 60
Number of participants with abnormal laboratory assessments during the study | Week 0 - Week 60
Number of participants with Clinically significant abnormal ECG results during the study | Week 0 - Week 60
WIN 378 Pharmacokinetics: concentration at trough [Ctrough] | Week 0 - Week 60
WIN 378 Pharmacokinetics: area under the concentration time curve [AUC] | Week 0 - Week 60
WIN 378 Pharmacokinetics: maximum observed concentration [Cmax]) | Week 0 - Week 60
Number of participants with positive anti-drug antibodies (ADA) during the study | Week 0 - Week 60

SECONDARY OUTCOMES:
Change from baseline in FeNO at Week 24 and Week 48 | Week 0 - Week 24, Week 48
Change from Baseline in Blood eosinophil count at Week 24 and Week 48 | Week 0 - Week 24, Week 48
Change in pre-BD and post-BD FEV1 at Week 24 and Week 48 | Week 0 - Week 24, Week 48
Change in pre-BD and post-BD forced vital capacity (FVC) at Week 24 and Week 48 | Week 0 - Week 24, Week 48
Annualized asthma exacerbation rate (AAER) over 48 weeks | Week 0 - Week 48
Annualized rate of severe asthma exacerbations over 48 weeks | Week 0 - Week 48
Time to first asthma exacerbation/severe asthma exacerbation over 48 weeks | Week 0 - Week 48
Proportion of participants with 1 or more asthma exacerbations/severe asthma exacerbations over 48 weeks | Week 0 - Week 48
Change from baseline in asthma symptoms (daytime and nighttime symptom frequency and severity, activity avoidance and limitation, asthma-related stress and fatigue as well as rescue asthma medication use) as measured by the Asthma Symptom Diary | Week 0 - Week 48
Change from baseline in Asthma Control Questionnaire (ACQ-6) at Week 48 | Week 0 - Week 48
Change from baseline in Asthma Quality of Life Questionnaire (Standardised) + 12 at Week 48 | Week 0 - Week 48
Change from baseline in European Quality of Life - 5 Dimensions 5 Level Version (EQ-5D-5L) at Week 48 | Week 0 - Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Omar Khwaja, MD, Study Director — Windward Bio
Locations (48):
- United States (17):
  - WB Contracted Clinical Research Site, Los Angeles, California
  - WB Contracted Clinical Research Site, San Jose, California
  - WB Contracted Clinical Research Site, Melbourne, Florida
  - WB Contracted Clinical Research Site, Miami, Florida
  - WB Contracted Clinical Research Site, White Marsh, Maryland
  - WB Contracted Clinical Research Site, Richfield, Minnesota
  - WB Contracted Clinical Research Site, St Louis, Missouri
  - WB Contracted Clinical Research Site, Bellevue, Nebraska
  - WB Contracted Clinical Research Site, Toledo, Ohio
  - WB Contracted Clinical Research Site, Edmond, Oklahoma
  - WB Contracted Clinical Research Site, Charleston, South Carolina
  - WB Contracted Clinical Research Site, Spartanburg, South Carolina
  - WB Contracted Clinical Research Site, Austin, Texas
  - WB Contracted Clinical Research Site, El Paso, Texas
  - WB Contracted Clinical Research Site, McKinney, Texas
  - WB Contracted Clinical Research Site, San Antonio, Texas
  - WB Contracted Clinical Research Site, Richmond, Virginia
- Australia (6):
  - WB Contracted Clinical Research Site, Brookvale, New South Wales
  - WB Contracted Clinical Research Site, Coffs Harbour, New South Wales
  - WB Contracted Clinical Research Site, Maroubra, New South Wales
  - WB Contracted Clinical Research Site, Miranda, New South Wales
  - WB Contracted Clinical Research Site, Wollongong, New South Wales
  - WB Contracted Clinical Research Site, North Altona, Victoria
- Bulgaria (4):
  - WB Contracted Clinical Research Site, Sofia, Grad Sofia
  - WB Contracted Clinical Research Site, Lovech, Lovech
  - WB Contracted Clinical Research Site, Rousse, Ruse
  - WB Contracted Clinical Research Site, Sofia, Sofia
- France (5):
  - WB Contracted Clinical Research Site, Pessac, Bordeaux
  - WB Contracted Clinical Research Site, Dijon, Côte-dOr
  - WB Contracted Clinical Research Site, Montpellier, Hérault
  - WB Contracted Clinical Research Site, La Tronche, Isère
  - WB Contracted Clinical Research Site, Nantes, Loire-Atlantique
- Germany (7):
  - WB Contracted Clinical Research Site, Berlin, Loire-Atlantique
  - WB Contracted Clinical Research Site, München, Loire-Atlantique
  - WB Contracted Clinical Research Site, Bendorf, Rhineland-Palatinate
  - WB Contracted Clinical Research Site, Darmstadt
  - WB Contracted Clinical Research Site, Frankfurt am Main
  - WB Contracted Clinical Research Site, Leipzig
  - WB Contracted Clinical Research Site, München
- Spain (7):
  - WB Contracted Clinical Research Site, Chiclana de la Frontera, Cádiz
  - WB Contracted Clinical Research Site, San Sebastián, Guipúzcoa
  - WB Contracted Clinical Research Site, Madrid, Madrid
  - WB Contracted Clinical Research Site, Pozuelo de Alarcón, Madrid
  - WB Contracted Clinical Research Site, Benalmádena, Málaga
  - WB Contracted Clinical Research Site, Málaga, Málaga
  - WB Contracted Clinical Research Site, Seville, Sevilla
- Sweden (2):
  - WB Contracted Clinical Research Site, Malmo, Skåne County
  - WB Contracted Clinical Research Site, Stockholm, Stockholm County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://windwardbio.com/